CLINICAL TRIAL: NCT06434701
Title: Severe COVID-19 Infection in Children Presenting to Emergency Departments in Israel and England: A Prospective Multicenter Study
Brief Title: Severe COVID-19 Infection in Children Presenting to EDs in Israel and England
Acronym: SPICE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hadassah Medical Organization (Other)
Collaborators: London North West Healthcare NHS Trust (Other)
Responsible Party: Principal Investigator, Itai Shavit, Chair, Division of Pediatrics, Hadassah Medical Center, Hadassah Medical Organization
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: SPICE-HMO-CTIL
Record Dates: First submitted 2024-05-21; First posted 2024-05-30 (Actual); Last update posted 2025-03-14 (Actual); Status verified 2025-03

CONDITIONS: COVID-19; Inflammatory Response
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Severe acute COVID-19 infection (Experimental): Nasopharyngeal swab sampling for COVID-19
  Interventions: Diagnostic Test: Nasopharyngeal swab sampling for COVID-19

INTERVENTIONS:
Diagnostic Test: Nasopharyngeal swab sampling for COVID-19 — The healthcare provider will gently insert the swab a short distance (1-1.5 cm for young children) into one nostril, reaching the back of the nasal cavity. The swab will then be gently rotated and rubbed for a few seconds to collect a sample of mucus. The same process may be repeated in the other nostril.

SUMMARY:
Even though the COVID-19 pandemic is no longer at its peak, the threat still lingers. Engaging in prospective surveillance studies will enable us to monitor the disease and prepare for any potential resurgence. COVID-19 surveillance studies are essential tools for policymakers to make informed decisions, allocate resources, and develop strategies to control the spread of the virus and protect public health.

The objective of this surveillance study is to prospectively assess in-hospital severe morbidity related to COVID-19 infection in children who present to the Pediatric Emergency Department (ED).

A prospective multicenter study will be conducted across eight EDs in Israel and five EDs in the United Kingdom. The study population will include children aged 16 years or younger with a severe acute COVID-19 infection. Confirmation of acute COVID-19 infection will be based on polymerase chain reaction nasopharyngeal swab testing. The study will also include patients diagnosed with multisystem inflammatory syndrome in children (MIS-C), as defined by the CDC.

ELIGIBILITY:
Inclusion Criteria:

1. SACI

   Patients aged 16 years or younger with a positive COVID-19 PCR nasopharyngeal swab testing or bronchoalveolar sample who meet the definition of SACI:
   * Receive oxygen via low-flow nasal cannula or oxygen mask, high-flow nasal cannula, bilevel or continuous positive airway pressure machine, mechanical ventilation, or extracorporeal membrane oxygenation (ECMO) Or
   * Admitted to ICU
2. MIS-C Patients aged 16 years or younger diagnosed with MIS-C

Ages: 0 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 500 (Estimated)
Dates: Start 2024-09-30 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Severe acute COVID-19 infection (SACI) | Up to 16 weeks
  The percentage of patients diagnosed with SACI among all patients admitted to the Emergency Department

SECONDARY OUTCOMES:
Administration of low-flow oxygen therapy via nasal cannula or face mask | Up to 12 weeks
  The percentage of COVID-19 patients treated with low-flow oxygen among all patients admitted to the Emergency Department
Administration of high-flow oxygen via nasal cannula (HFNC), or administration of oxygen via bilevel or continuous positive airway pressure (CPAP) machine | Up to 12 weeks
  The percentage of COVID-19 patients treated with HFNC or CPAP among all patients admitted to the Emergency Department
Treatment with mechanical ventilation | Up to 12 weeks
  The percentage of COVID-19 patients treated with mechanical ventilation among all patients admitted to the Emergency Department
Treatment with extracorporeal membrane oxygenation (ECMO) | Up to 8 weeks
  The percentage of COVID-19 patients treated with ECMO among all patients admitted to the Emergency Department
Treatment with vasopressor support | Up to 8 weeks
  The percentage of COVID-19 patients treated with vasopressor support among all patients admitted to the Emergency Department
Length of ICU stay | Up to 16 weeks
  Mean duration of ICU stay for patients admitted with COVID-19
Length of hospital stay | Up to 24 weeks
  Mean duration of hospital stay for patients admitted with COVID-19

CONTACTS AND LOCATIONS:
Locations (6):
- Israel (6):
  - Haemek Medical Center, Afula
  - Soroka Medical Center, Beersheba
  - Hadassah Medical Center, Jerusalem
  - Shaare Zedek Medical Center, Jerusalem
  - Meir Medical Center, Kfar Saba
  - Sheba Medical Center, Tel Litwinsky

IPD SHARING:
Plan to Share IPD: No